CLINICAL TRIAL: NCT01139099
Title: Department of Psychiatry of NTUH Yun-Lin Branch
Brief Title: The Evaluation of Therapeutic Efficacy on the Integrated Group Psychotherapy for Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201003068R
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm (Other): There is no arm in this study.
  Interventions: Behavioral: Group Psychotherapy

INTERVENTIONS:
Behavioral: Group Psychotherapy — integrated group psychotherapy, including the interpersonal and cognitive group therapy

SUMMARY:
Although the patients with schizophrenia can be treated with new generation of antipsychotics medication, additional approaches are necessary to improve schizophrenics' cognitive functions, interpersonal relationships as well as social adjustment. When some of patients return to community, they expose to practical pressure that contribute to worsen and relapse of disease. That further damages patient's cognitive functions. Integrated Psychological Therapy(IPT) on treating schizophrenia has dramatic improvement in recent years; it has formed structured treatment gradually on relieving illusion, hallucination as well as negative symptoms. This study aims at conducting 12-week structured IPT group therapy. The intended subjects are patients, met with DSM-Ⅳ-TR diagnosis of schizophrenia, from community, outpatient and inpatient service. The overall treatments are designed to provide 1-2 hours weekly group therapy which focuses on relieving illusions, hallucination, and negative symptoms. Patients' cognitive functions, ability of emotional adjustment and interpersonal relationship would be evaluated in pre-test and post-test to indicate whether the significant difference exists. There is a controlled group, in which patients who still receive treatment as usual (TAU). The study also compares the evaluation results between IPT group and TAU group, hoping to develop the therapeutic framework for Taiwan people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia,
* can concentrate in group for 30 minutes.

Exclusion Criteria:

* substance abuse (alcohol, illegal medication),
* self harm history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
re-hospitalization rate | after 3 months of the group psychotherapy
  acute symptom relapse and needed to be admitted to the acute ward

SECONDARY OUTCOMES:
Cognitive functions, ability of emotional adjustment, and interpersonal relationship | 12 months of the group tpsychotherapy
  The tests of psychiatric symptoms, cognitive test, anxiety, depression, interpsersonal skill, and emotional adjustment Add Secondary Outcome Measure:The Positive and Negative Syndrome Scale, Beck depression scale, Beck anxiety scale, Beck suicial ideation scale, Cognitive tests (visual spatial test), CPT-IP for attention test
The Positive and Negative Syndrome Scale, Beck depression scale, Beck anxiety scale, Beck suicial ideation scale, Cognitive tests (visual spatial test), CPT-IP for attention test | 12 months of the group psychotherapy
  The Positive and Negative Syndrome Scale for psychiatric symptoms, Beck depression scale for depression symptoms, Beck anxiety scale for anxiety symptoms, Beck suicial ideation scale for suicidal ideation evalution Cognitive tests (visual spatial test), CPT-IP for attention test for cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ren Chang, MD, Study Director — Department of Psychiatry in National Taiwan University Hospital Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital Yun-Lin Branch, Douliu, Taiwan, Taiwan